CLINICAL TRIAL: NCT01741714
Title: Is Chiropractic Spinal Manipulative Therapy an Efficient Treatment Option for Migraine? A Randomized Controlled Clinical Trial
Brief Title: Is Chiropractic Spinal Manipulative Therapy an Efficient Treatment Option for Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Collaborators: Norwegian Foundation for Health and Rehabilitation (Other); Norwegian Chiropractic Association (Unknown)
Responsible Party: Principal Investigator, Aleksander Chaibi, PhD student, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Migraine-K34KSF-AHUS; 2829002 (Other Grant/Funding Number: 2829002)
Record Dates: First submitted 2012-12-02; First posted 2012-12-05 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Migraine With Aura; Migraine Without Aura
MeSH Terms: conditions — Migraine with Aura; Migraine without Aura

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Chiropractic Spinal Manipulative Therapy (Active Comparator): Active chiropractic spinal manipulative treatment
  Interventions: Other: Chiropractic spinal manipulative therapy
- Sham manipulation (Sham Comparator): Sham chiropractic manipulative therapy
  Interventions: Other: Sham chiropractic manipulative therapy
- Control group (No Intervention): No intervention, follow headache diary

INTERVENTIONS:
Other: Sham chiropractic manipulative therapy — Sham manipulation
  Arms: Sham manipulation
Other: Chiropractic spinal manipulative therapy — Chiropractic spinal manipulative therapy
  Arms: Chiropractic Spinal Manipulative Therapy

SUMMARY:
This study will highlight and validate chiropractic spinal manipulative therapy (CSMT) for migraine. If the method proves to be effective, it will provide a new non-pharmacological treatment option for migraine. This is especially important since some migraineurs do not tolerate acute and/or prophylactic medicine, due to side effects or contraindications due to comorbidity of other diseases while others do not have effect. Thus, alternative treatment options are warranted. The applied methodology of the study will aim towards the highest possible research standards. This international study is a collaboration between Akershus University Hospital, University of Oslo (UiO), Norway and Macquarie University, Australia. The multidisciplinary professional backgrounds are physiotherapy, chiropractic and medicine. By increasing the methodological quality of the investigators research to a very high level, the investigators see the method to work as a guide to increase the quality of chiropractic research in the future, as previous randomized clinical trials (RCTs) of migraine used methodology showing room for improvement.

DETAILED DESCRIPTION:
Migraine is characterized by a unilateral pulsating moderate/severe headache which is aggravated by routine physical activity, and is accompanied by photo- and/or phonophobia, nausea and sometimes vomiting. Migraine exists in two forms, migraine without aura (MO) and migraine with aura (MA). Aura is reversible neurological disturbances of the vision, sensory and/or speech, which occur prior to the headache. The aura symptoms show intra-individual variations. The origin of migraine pain is still debated, since the origin of painful impulses in the trigeminal nerve is still uncertain. Some argues for central and other argues for peripheral mechanisms. Extracranial pain sensitive structures include skin, muscles, arteries, periosteum and joints. The skin is sensitive to all usual forms of pain stimuli, while especially temporal and neck muscles may be sources for pain and tenderness in migraine. Similarly is the frontal supraorbital, superficial temporal, posterior and occipital arteries sensitive to pain. It has been hypothesize that CSMT might relieve migraine due to stimulation of different mechanoreceptors in the neck such as the zygapophyseal joints, intervertebral discs and neck muscles. Numerous studies of manipulations have been conducted, but all had one or more methodological shortcomings, i.e. failure to specify diagnostic criteria, inadequate or no randomization procedure, lack of control, lack of patient blinding, lack of specified primary and secondary end points and shortcomings of statistical evaluation of the results. A few RCTs suggest that CSMT using diversified technique is an effective therapy for migraine. The diversified technique is used by 91% of chiropractors, and include a collections of procedures, hence the name diversified. It focuses on inter-segmental pretension (soft tissue tension) prior to the delivery of high velocity low amplitude (HVLA) adjustment. The Gonstead method is used by 59% of chiropractors and is also based on HVLA, but a major difference is the minimal usage of rotation in all adjustments in contrast to the diversified technique. The Gonstead method is considered safe, since severe adverse reactions have not been encountered. No studies have previously investigated the efficacy of the Gonstead method for migraine, although research in other CSMT modalities has been recommended.

Study hypothesis CSMT using the Gonstead method reduces days with migraine by at least 25% as compared to placebo (sham manipulation, i.e. broad non-specific contact, non-directional, low velocity and low amplitude) and no intervention (control group).

The RCT is single blinded, placebo-controlled trial of CSMT using the Gonstead method vs. sham manipulation and control group. If the treatment shows to be effective, the participants whom receive sham manipulation or control will be offered true intervention after the follow-up period and free of charge. This study will follow the recommendations set by the clinical trial guidelines from the IHS, while the methodological quality control will in general follow previous suggested criteria and the CONSORT statements.

Patients will be recruited through Akershus University Hospital, Norway as well as through media advertising in Akershus and Oslo County. The diagnoses are set by a chiropractor and a neurologist with experience in headache. In accordance with good clinical practice, all patients will receive written and oral information about the project and will be informed about the harms and benefits as well as adverse reaction of the intervention. A total of 90 participants need to be recruited to the clinical trial.

The clinical trials consist of three stages: Run-in, intervention (treatment) and follow-up.

One month of baseline data collection where participants will fill-in a diagnostic headache diary. Baseline demographics and clinical characteristics will be presented in tables with mean and standard deviation (SD) for each group.

As age and genders may plays a role, participants will be subdivided into four subgroups by age and gender prior to the concealed group allocation and restricted randomization by drawing prepared sealed lots. Each lot includes three different interventions, i.e active treatment, sham manipulation and control group. The first three participants will draw from the same lot until all three interventions are used. The next lot with three interventions is then followed by the next three participants; each participant will only receive one intervention.

The RCT will be conducted by an experienced chiropractor. Active treatment consists of CSMT using the Gonstead method. A specific contact, high velocity, low amplitude, short lever, with no recoil post adjustment directed to spinal biomechanical dysfunction diagnosed by standard chiropractic tests.

Follow-up at 3, 6 and 12 months post-treatment. During this period participants continue to fill in a diagnostic headache diary. The control group will also be included in this phase of the study.

The data will be analyzed with SPSS using standard statistical techniques.

The investigators based the calculation of sample size on migraine days from recent group comparison studies of topiramate. The investigators calculated that a sample size of 16 patients was required in each group to detect a difference in mean reduction in monthly migraine headache days of 2.5 with 80% power, with p=0.05 as level of significance, and assuming a common SD of 2.5 for active treatment and broad-based treatment groups.

Insurance is through "The Norwegian System of Compensation to Patients" (NPE) which is an independent national body, set up to process compensation claims from patients who have suffered an injury as a result of treatment under the Norwegian health service.

The Regional Committee for Medical Research Ethics (REK) in Norway and Norwegian Social Science Data Services approved the full PhD research protocol. The declaration of helsinski is followed.

ELIGIBILITY:
Inclusion Criteria:

* Migraine according to the diagnostic criteria of the ICHD-II (8)
* At least one migraine attack per month
* Age 18-70 years

Exclusion Criteria:

* Contraindication to spinal manipulation
* Chiropractic treatment within the last 12 months
* Radiculopathy
* Depression
* Pregnancy
* Participants whom become pregnant during the migraine trial will also be excluded from analysis from the time of pregnancy
* Participants who change their prophylactic medical regime for headaches will be excluded in the analysis from the time of change

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2013-02; Primary Completion 2015-03 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Number og headache days | Change from baseline to post-treatment, 3, 6, 12 months follow-up
  1. 25% reduction in number of headache days between active treatment and sham.
  2. 25% reduction in number of headache days between active treatment and control group.

SECONDARY OUTCOMES:
Headache duration | Change from baseline to post-treatment, 3, 6, 12 months follow-up
  1. 25% reduction in headache duration in hours between active treatment and sham.
  2. 25% reduction in headache duration in hours between active treatment and control group.
Self reported VAS | Change from baseline to post-treatment, 3, 6, 12 months follow-up
  1. 25% self-reported improvement on VAS between active treatment and sham.
  2. 25% self-reported improvement on VAS between active treatment and control group.
Headache index | Change from baseline to post-treatment, 3, 6, 12 months follow-up
  1. 25% reduction in headache index (frequency x duration x intensity) between active treatment and sham.
  2. 25% reduction in headache index between active treatment and control group.
Headache medication | Change from baseline to post-treatment, 3, 6, 12 months follow-up
  1. 50% reduction in headache medication between active treatment and sham.
  2. 50% reduction in headache medication between active treatment and control group.

OTHER OUTCOMES:
Sub analysis on x-ray findings | Pre-treatment
  As there are no validated x-ray assessment forms a descriptive sub-analysis will be done on participants with structural deformities vs. normal x-ray findings. Structural deformities include postural assessment, joint and disc integrity, vertebral misalignments and ruling out pathology prior to CSMT.

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Russell, Professor, Study Director — Head and Neck Research Group, Research Centre, Akershus University Hospital
Locations (1):
- Research Centre, Akershus University Hospital, Lørenskog, Norway

REFERENCES:
- [Background] Chaibi A, Tuchin PJ, Russell MB. Manual therapies for migraine: a systematic review. J Headache Pain. 2011 Apr;12(2):127-33. doi: 10.1007/s10194-011-0296-6. Epub 2011 Feb 5. PMID 21298314
- [Background] Chaibi A, Saltyte Benth J, Tuchin PJ, Russell MB. Chiropractic spinal manipulative therapy for migraine: a study protocol of a single-blinded placebo-controlled randomised clinical trial. BMJ Open. 2015 Nov 19;5(11):e008095. doi: 10.1136/bmjopen-2015-008095. PMID 26586317
- [Result] Chaibi A, Benth JS, Tuchin PJ, Russell MB. Chiropractic spinal manipulative therapy for migraine: a three-armed, single-blinded, placebo, randomized controlled trial. Eur J Neurol. 2017 Jan;24(1):143-153. doi: 10.1111/ene.13166. Epub 2016 Oct 2. PMID 27696633
- [Result] Chaibi A, Saltyte Benth J, Bjorn Russell M. Validation of Placebo in a Manual Therapy Randomized Controlled Trial. Sci Rep. 2015 Jul 6;5:11774. doi: 10.1038/srep11774. PMID 26145718
- [Result] Chaibi A, Benth JS, Tuchin PJ, Russell MB. Adverse events in a chiropractic spinal manipulative therapy single-blinded, placebo, randomized controlled trial for migraineurs. Musculoskelet Sci Pract. 2017 Jun;29:66-71. doi: 10.1016/j.msksp.2017.03.003. Epub 2017 Mar 14. PMID 28324697